CLINICAL TRIAL: NCT01415388
Title: A Double-blind, Randomized, Multi-centre, Placebo-controlled Study to Investigate the Effects of Superba(TM) Krill Oil on Fasting Serum Triglycerides
Brief Title: Study to Investigate the Effects of Krill Oil on Fasting Serum Triglycerides
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aker BioMarine Human Ingredients AS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CHSI 1102-16
Record Dates: First submitted 2011-08-10; First posted 2011-08-12 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
Keywords: Maintenance of normal blood triglyceride levels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Krill Oil — 4 Capsules twice daily providing 0 (placebo), 0.5, 1.0, 2.0, or 4.0 g krill oil/day for a period of 12 weeks
  Other Names: Superba(TM) Krill Oil

SUMMARY:
The purpose of this study is to assess the effect of 12 weeks of daily supplementation with Superba(TM) Krill Oil on fasting serum triglyceride levels and omega-3 index in subjects whose habitual fatty fish and seafood intake is low and who have borderline high or high fasting serum triglyceride levels.

ELIGIBILITY:
Inclusion Criteria(not limited to):

* General good health with no existing co-morbidities
* Body mass index (BMI) less than 35 kg/m²
* Borderline high or high fasting serum triglycerides
* Clinically normal findings for hematology, clinical chemistry, and urinalysis
* Be willing to maintain dietary habits and physical activity levels throughout the trial period (next 4 months)
* Have a low habitual consumption of fatty fish and seafood, defined as a frequency of twice per month or less

Exclusion Criteria (not limited to):

* Familial hypercholesterolemia or severely high total cholesterol levels
* History or presence of significant cardiovascular disease or co-morbidities
* Known allergy to crustaceans (shellfish)
* Bleeding disorders
* Disturbed absorption due to changes in the gastrointestinal tract
* Participation in a clinical trial with an investigational product within 30 days before screening
* Present or recent use (within 3 months of screening or the first screening visit, if applicable) of any medication which is a known lipid modifying agent or any dietary supplements that affect the level of blood cholesterol and triglycerides
* Current or recent diet, which in the opinion of the Investigator, deviates from a normal diet (e.g., vegetarians may be acceptable, vegans are not acceptable)
* Female patients that are pregnant or nursing or females of childbearing potential who are not on a method of birth control acceptable to the Investigator during treatment
* Patients with known coagulopathy or receiving anticoagulant therapy or co-morbidity that would interfere with the study results
* Frequency of fatty fish and/or seafood consumption is greater than twice per month
* Present or recent use of any long-chain omega-3 fatty acid supplement
* Peri-menopausal women or post-menopausal women taking hormone replacement therapy
* Patients who test positive for human immunodeficiency virus (HIV) or hepatitis B or C
* Systolic blood pressure greater than 159 mmHg or diastolic blood pressure greater than 99 mmHg or use of anti-hypertensive medication
* Diabetic subjects
* Staff of Cetero Research

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Change in fasting serum triglycerides | Baseline (Day 1) and at Day 85

SECONDARY OUTCOMES:
Omega-3 index | At Days 1, 42, and 85

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cetero Research, Saint Charles, Missouri
  - Cetero Research, Fargo, North Dakota